CLINICAL TRIAL: NCT02948270
Title: Communication in Adolescents With ADHD
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rosemary Tannock, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000026311
Record Dates: First submitted 2015-05-25; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents with ADHD: Adolescents who met diagnostic criteria in previous clinical/research assessment are invited to come back to SickKids to participate (ages 13-17)
- Adolescents without ADHD: Adolescent controls (ages 13-17) are tested through local high schools

SUMMARY:
The interpersonal problems of adolescents with ADHD may be the most debilitating aspect of their psychopathologic behaviour. This being said, the investigators still do not have a clear understanding of why it is the case that individuals with ADHD have such impaired social and communicative competence. In particular, research has not identified whether the communicative difficulties stems from deficits in taking the perspective of a communicative partner, or in being able to make use of this information in a systematic way. This study will compare adolescents with ADHD to adolescents not diagnosed with ADHD and their performance on a number of social inference and communication tests. This study hypothesizes that persons with ADHD will not perform as effectively as control participants on the social inference and communication tests, and will evidence lower WM score. As well, this study hypothesizes that a working memory/cognitive load task will impede performance on certain social inference and communication tests to a greater extent in the ADHD population than in the control group.

DETAILED DESCRIPTION:
The first objective of this project is to examine whether individuals with ADHD symptoms are less able than their non-ADHD counterparts to use the perspective of their conversational partner, a deficiency which in turn contributes to increased difficulty in more complex communicative contexts.

The second objective is to assess the degree to which communicative difficulties stem from the core cognitive deficits faced by individuals with ADHD. Only recently has the developmental literature uncovered the relationship between cognitive skills and communicative perspective-taking. That is, children who have more proficient inhibition are better able to suppress their own perspective in order to take into account the perspective of a conversational partner (Nilsen & Graham, 2009). Furthermore, working memory skills have been found to relate to children's ability to understand the intentions of speakers who use figurative language (e.g., Filippova & Astington, 2008).Thus, it may be that a weakness in inhibition and working memory (over and above possible weakness in their mentalizing skills) prevents children with ADHD from using the perspective of their conversational partner during communicative interactions.

General research questions: Are adolescents with ADHD less able to appreciate the perspective of conversational partners? Does this relate to their core executive deficits?

Specific Research Questions Summary:

1. Do adolescents with ADHD show less social inference ability? Is this ability exacerbated by increased cognitive demands (e.g., working memory)?
2. Do adolescents with ADHD show less communicative perspective-taking? Is this related to their inhibitory control skills?
3. Do adolescents with ADHD overestimate the clarity of their intended messages in texts? Is this 'overestimation' more closely related to difficulties with appreciating 'common ground' when constructing text messages?
4. Do adolescents with ADHD conflate their own knowledge with that of a listener in third-person perspective tasks? Is this related to IC / WM?

   Other questions that can be examined in the proposed study, but not outlined specifically here:
5. Do adolescents that show difficulty on the communicative perspective-taking tasks show worse overall social competence? (self/parent report)
6. Is the social outcome worse for girls than boys, due to the more intimate social milieu of girls compared to relatively loose social networks of adolescent boys? (e.g., Ohan & Honston, 2007).
7. Do self-reported EF difficulties relate to actual EF performance? Do self-reported EF difficulties relate to performance on the perspective-taking tasks?

Proposed procedure:

* Adolescents who met diagnostic criteria in previous clinical/research assessment are invited to come back to SickKids to participate in research study (ages 13-17)
* Adolescent controls are tested through local high schools

Task summary:

Social / communicative perspective-taking tasks:

* The Awareness of Social Inference Test (TASIT, McDonald et al., 2002)
* Without working memory load (10 min)
* With working memory load (10 min)
* Computerized Perspective-taking (Apperly) (10-15 min)
* Texting task (similar to Kruger et al., ) (15 min)
* Story Vignette task (15 min)

Executive function tasks:

Inhibitory Control measures:

* Stroop (5 min)
* Stop Signal (15 min)

Working Memory measures:

* Sentence span (10 min)
* WRAML finger windows (10 min)

Report measures:

* The SNAP-IV Teacher and Parent Rating Scale
* Social Skills Improvement System (SSIS, Gresham & Elliot, 2007) parent report 3-18
* Strengths and Difficulties Questionnaire (SDQ) Adolescent:
* Behavior Rating Inventory of Executive Functioning (BRIEF) SR 11-18 years
* Social Skills Improvement System (SSIS, Gresham & Elliot, 2007) student report 13-18
* Strengths and Difficulties Questionnaire (SDQ) Parent

Information required from past adolescents' past participation:

* ADHD diagnostic status
* Any other diagnoses (e.g., LD / ODD)
* Cognitive level (FSIQ, VCI, PRI)

ELIGIBILITY:
Inclusion Criteria:

* ADHD

Exclusion Criteria:

* Other mental health diagnoses, such as ASD.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents from ages 14 to 17 with and without ADHD
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Use of perspective in conversation | Up to 3 hours during assessment

SECONDARY OUTCOMES:
The degree to which communicative difficulties stem from the core cognitive deficits | Up to 3 hours during assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ferguson, MD, Principal Investigator — The Hospital for Sick Children; Rosemary Tannock, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No